CLINICAL TRIAL: NCT01718223
Title: A Pilot Study of Interstitial Photodynamic Therapy for Recurrent Squamous Cell Carcinoma of the Oropharynx and Oral Cavity
Brief Title: Photodynamic Therapy Using Temoporfin Before Surgery in Treating Patients With Recurrent Oral Cavity or Oropharyngeal Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: implementation issues
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Biolitec Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 217512; NCI-2012-01879 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Stage I Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage I Squamous Cell Carcinoma of the Oropharynx; Stage I Verrucous Carcinoma of the Oral Cavity; Stage II Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage II Squamous Cell Carcinoma of the Oropharynx; Stage II Verrucous Carcinoma of the Oral Cavity; Tongue Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; temoporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (interstitial photodynamic therapy using temoporfin) (Experimental): Patients receive temoporfin IV over at least 6 minutes on day 1 and undergo interstitial photodynamic therapy on day 3. Within 4-6 weeks, patients undergo surgical resection.
  Interventions: Drug: photodynamic therapy; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis; Drug: temoporfin

INTERVENTIONS:
Drug: photodynamic therapy — Undergo interstitial photodynamic therapy using temoporfin
  Other Names: Light Infusion Therapy™; PDT; therapy, photodynamic
Procedure: therapeutic conventional surgery — Undergo surgical resection
Other: laboratory biomarker analysis — Correlative studies
Drug: temoporfin — Undergo interstitial photodynamic therapy using temoporfin
  Other Names: Foscan; m-tetrahydroxyphenyl-chlorin; mTHPC

SUMMARY:
This pilot clinical trial studies photodynamic therapy using temoporfin before surgery in treating patients with recurrent oral cavity or oropharyngeal cancer. Photodynamic therapy uses a drug, such as temoporfin, that is absorbed by tumor cells. The drug becomes active when it is exposed to light. When the drug is active, tumor cells are killed. Giving photodynamic therapy using temoporfin before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the toxicity of dose regimen using the Cancer Therapy Evaluation Program (CTEP) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE version 4.0).

SECONDARY OBJECTIVES:

I. Quantify the relationship between the measured intra-tumor light dose and the pathological tumor response.

TERTIARY OBJECTIVES:

I. Simulate light dose distribution within the treated tumor. II. Immune markers.

OUTLINE:

Patients receive temoporfin intravenously (IV) over at least 6 minutes on day 1 and undergo interstitial photodynamic therapy on day 3. Within 4-6 weeks, patients undergo surgical resection.

After completion of study treatment, patients are followed for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Histologically confirmed recurrent or T2/T3/T4 squamous cell carcinoma of the oropharynx or oral cavity that are amenable to surgery
* Tumor accessible for unrestricted illumination for interstitial photodynamic therapy (PDT) (accessibility as determined by the physician)
* Life expectancy of at least 6 months in the judgment of the physician
* Blood urea nitrogen (BUN) =< upper limit of normal (ULN)
* White blood count > 3,000 per microliter or
* Absolute neutrophil count (ANC) > 1500 per microliter
* Serum calcium within normal limits; note: serum calcium will be corrected for low albumin, if necessary
* Subjects of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Subject or legal representative must understand the investigational nature of this study and sign an Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Subjects who have had radiotherapy within the last 3 months
* Subjects with known brain metastases should be excluded from this clinical trial
* Tumor invading a major blood vessel (such as the carotid artery)
* Tumor invading the skull base
* Subjects with ophthalmic disease
* Tumor is not clearly shown on an imaging scan/location and extension of tumor that precludes effective PDT, in the judgment of the primary investigator (PI)
* Location and extension of the tumor precludes an effective interstitial photodynamic therapy (iPDT)
* Patients with known hypersensitivity to porphyrins or with porphyria
* Has distant metastasis that decreases life expectancy to less than 6 months
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing female subjects
* Unwilling or unable to follow protocol requirements and the light exposure precautions
* Any condition which in the investigator's opinion deems the subject an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events, graded according to NCI CTCAE version 4.0 | Up to 30 days after surgical resection
  The frequency of toxicities will be tabulated by grade.

SECONDARY OUTCOMES:
Light dose-volume histograms (DVH), defined as the overall light dose (joules) that was delivered to the tumor volume throughout the therapy with the light dosimetry system | Day 3
Ratio of the viable/nonviable tissue in the resected tumor, ex vivo | Up to 6 weeks
  The area of viable and necrotic tumor will be measured by the number of field of view (1 FOV = 0.196 mm^2), microscopic area using a 40x objective.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Arshad, MD, Principal Investigator — Roswell Park Cancer Institute